CLINICAL TRIAL: NCT00002674
Title: CYTOREDUCTIVE CHEMOTHERAPY WITH MITOXANTRONE, CYTOSINE ARABINOSIDE AND ETOPOSIDE FOLLOWED BY RECOMBINANT HUMAN G-CSF FOR MOBILIZATION OF PERIPHERAL BLOOD STEM CELLS IN PATIENTS WITH CHRONIC MYELOID LEUKEMIA
Brief Title: Combination Chemotherapy Followed by Peripheral Stem Cell Transplantation in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 928.00; FHCRC-928.00; NCI-H95-0705; CDR0000064310 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-08-23 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Filgrastim; Cytarabine; Etoposide; Hydroxyurea; Mitoxantrone; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: cytarabine
Drug: etoposide
Drug: hydroxyurea
Drug: mitoxantrone hydrochloride
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy used to kill cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by G-CSF and peripheral stem cell transplantation in treating patients with chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of MCE (mitoxantrone/cytarabine/etoposide) followed by granulocyte colony-stimulating factor to mobilize peripheral blood stem cells (PBSC) in patients with chronic myeloid leukemia (CML). II. Evaluate the toxicity of this regimen. III. Evaluate the cytoreductive effects of this regimen in CML as determined by the ability to mobilize Philadelphia chromosome-negative PBSC. IV. Assess the time of peak CD34+ and CD34+/CD38- cell concentrations in the peripheral blood of patients treated with this regimen.

OUTLINE: The following acronyms are used: ARA-C Cytarabine, NSC-63878 DHAD Mitoxantrone, NSC-301739 G-CSF Granulocyte Colony-Stimulating Factor (source not specified) HU Hydroxyurea, NSC-32065 MCE DHAD/ARA-C/VP-16 VP-16 Etoposide, NSC-141540 Single-Agent Cytoreduction followed by 3-Drug Combination Chemotherapy/Stem Cell Mobilization. HU; followed by MCE; G-CSF.

PROJECTED ACCRUAL: 30 patients will be entered over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Philadelphia chromosome-positive chronic myeloid leukemia (CML) in chronic or accelerated phase Ineligible for allograft protocols or no available HLA-matched sibling marrow donor No patients under age 55 who have consented to unrelated donor search unless: Search unsuccessful for 6 months and unlikely a donor will be found Transplant from an unrelated donor declined No history of CML blast crisis No grade III/IV myelofibrosis

PATIENT CHARACTERISTICS: Age: Over 17 to under 66 Performance status: Not specified Life expectancy: No limitations from disease other than leukemia Other: No hepatic, renal, pulmonary, or cardiac dysfunction that would preclude transplant preparative regimen No HIV antibody No active infection

PRIOR CONCURRENT THERAPY: At least 1 month since interferon

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1994-10; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona A. Holmberg, MD, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States